CLINICAL TRIAL: NCT03225066
Title: A Prospective, Randomized, Multicenter, Self-controlled, Blinded Trial on the Efficacy and Safety of Poly-L-lactic Acid - SCULPTRA - for the Treatment of Corporal Skin Flaccidity.
Brief Title: Efficacy and Safety of Poly-L-lactic Acid
Acronym: Sculptra
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma Brasil Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR.16.001
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2017-08

CONDITIONS: Flaccidity, Muscle
MeSH Terms: conditions — Muscle Hypotonia

STUDY DESIGN:
Intervention Model Description: The study sample will be stratified to include 50% of subjects, who will receive Sculptra treatment on the antero-medial side of the arms and approximately 50% of subjects, who will receive Sculptra treatment in the gluteal area, in order to exploratory analyzes by subgroup.
  During the study, the subjects should come to the research site up to nine times: one for the screening/inclusion visit (SV), three treatment visits (TVs) for Side 1 (from 1 to 14 days after SV, and from 1 to 2 months after first session), three TVs for Side 2 (4, 5 and 6 months after the first S1 treatment session), one follow-up visit (FUV), 6 months after the first S2 treatment session) and a final visit (FV) (12 months after the first S1 session). After 4 months of the first treatment we will compare the results between the first treated side and non-treated side.
Masking Description: P.S. To assess the efficacy of Sculptra, via adapted Global Aesthetic Improvement Scale score determined by blind evaluator (Outcomes assessor ), in the treatment of skin flaccidity on the anteromedial region of arm and gluteal region, 4 months after initiating the treatment, based on the assessment of the corporal side randomized to be the first to receive treatment. I input as NO MASKING because appears ERROR when I included Outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Poly-L-Lactic Acid - Sculptra (Experimental): Each area will be treated with a dose contained in a vial of Sculptra®. For conducting the study, six vials of the product will be available per subject, and one vial will be used in each session with up to maximum a total volume of 16mL per treated area. It will be 3 session with interval of 1 month in total.
  Interventions: Device: Poly-L-lactic acid - Sculptra

INTERVENTIONS:
Device: Poly-L-lactic acid - Sculptra — Participants using Sculptra - Poly-L-lactic acid 3 sessions in the first side and 3 sessions on the second side

SUMMARY:
This study aims to assess efficacy and safety of Sculptra in the treatment of skin flaccidity in selected areas - arms, anteromedial region, and gluteal regions. To assess the efficacy of Sculptra®, via adapted Global Aesthetic Improvement Scale -GAIS- score determined by blind evaluator, in the treatment of skin flaccidity on the anteromedial region of arm and gluteal region, 4 months after initiating the treatment, based on the assessment of the corporal side randomized to be the first to receive treatment . Considering as an alternative hypothesis of interest a 70% value of the subjects the treated side would have higher GAIS than the untreated side.

DETAILED DESCRIPTION:
Ethical and General considerations regarding the study conduction: This study protocol will be reviewed and approved by appropriate IEC/IRB prior to the initiation of the study.

Clinical monitoring: Study conduction will be closely monitored by Galderma representatives, following GCP regulations, applicable standard operating procedures, guides and local regulations.

Data Management: Data may be audited by Galderma Quality Assurance Department and/or CRO prior to or after results of the first statistical analysis on the primary discretion.

Quality assurance, auditing and Inspection: The study will be carried out under the sponsorship of Galderma in accordance with all local and federal regulations, as well as ICH guidelines. Audits and inspections at the research site may be conducted by Galderma representatives or local authorities. All aspects in any study step can be audited by Galderma Quality Assurance / CRO and, as a result, a certificate stating this will be provided.

ELIGIBILITY:
Inclusion Criteria:

1. Female;
2. Age between 35 and 60 years (including 60 years);
3. Indication for treatment of bilateral skin flaccidity of at least one of two corporal areas candidate for treatment (arms [anteromedial region] or gluteal regions);
4. Mild to moderate flaccidity in the area to be treated, according to investigator's assessment and in accordance with appropriated flaccidity scales for corporal region to be treated;
5. Subjects who understood and signed the Informed Consent Form (ICF) when entering the study, before performing any investigational procedure

Exclusion Criteria:

1. Prior use (<1 year) or planning to use any other aesthetic treatment in the corporal area of interest for study, such as radiofrequency, cryolipolysis;
2. History of liposuction, plastic surgery and / or corrective plastic surgery in the area of the body of interest for the study (arms or gluteal region);
3. History (<1year) of treatment with Sculptra in other corporal area, area without interest for study;
4. History of Sculptra treatment in the area of the body of interest for the study (arms or gluteal region);
5. Any type of comorbidity or clinical condition that, at investigator s discretion, could interfere with study assessments;
6. Using or planning to initiate restrictive diets (at investigator s discretion);
7. Using or planning to initiate use of supplements for weight loss;
8. Diabetes mellitus type 1 or type 2;
9. Autoimmune diseases, collagenosis, decompensated endocrine diseases or any disease that, at investigator's discretion, could interfere with study assessments;
10. Using or have used within 3 months drugs such as corticosteroids, immunosuppressants or others collagen-production inhibitors;
11. Initiated use of hormones or change in dose of hormonal replacement therapy within 3 months;
12. Practices regularly or intend to practice during the study high-performance or impact physical activities, such as weight lifting, marathon, triathlon;
13. Pregnant or breastfeeding, or wishes to get pregnant within the next 18 months, or refuses to use appropriate contraceptive method (in case of women of childbearing potential).

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Assess the aesthetic effect through photographs via GAIS score determined by blind evaluator | 4 months after starting Side 1 treatment
  To see the percentage of research subjects, to which the blind evaluator assigned a Global Aesthetic Improvement Scale score (GAIS) score higher to Side 1 than the corporal side which will be the second to receive treatment (Side 2), 4 months after starting Side 1 treatment.

SECONDARY OUTCOMES:
Assess the frequency with which the blind evaluators identified correctly Side 1, 4 months after initiating treatment on Side 1 through photographs. | 4 months after starting Side 1 treatment
  1. Percentage of evaluators identifying correctly the first treated side, 4 months after initiating treatment on Side 1.
Assess efficacy of Sculptra in the treatment of skin flaccidity via GAIS score determined by the investigator. | 4, 6 and 12 months after starting side 1 treatment and 6 and 8 months after starting side 2
  3.1. Mean GAIS score assigned by the investigator to Side 1, 4 months after initiating treatment.
  3.2. Mean GAIS score assigned by the investigator to Side 1, 6 months after initiating treatment.
  3.3. Mean GAIS score assigned by the investigator to Side 1, 12 months after initiating treatment.
  3.4. Mean GAIS score assigned by the investigator to Side 2, 6 months after initiating treatment.
  3.5. Mean GAIS score assigned by the investigator to Side 2, 8 months after initiating treatment.
To assess the aesthetic effect of Sculptra in the skin flaccidity treatment, treatment, via GAIS score determined by the research subject. | 4, 6 and 12 months after initiating side 1 as well as 6 and 8 months after initiating side 2 treatment
  4.1. Mean GAIS score assigned by the research subject to Side1, 4 months after initiating treatment.
  4.2. Mean GAIS score assigned by the female subject to Side1, 6 months after initiating treatment.
  4.3. Mean GAIS score assigned by the female subject to Side1, 12 months after initiating treatment.
  4.4. Mean GAIS score assigned by the female subject to Side2, 6 months after initiating treatment.
  4.5. Mean GAIS score assigned by the female subject to Side2, 8 months after initiating treatment.
To assess aesthetic effect of Sculptra on skin flaccidity via GAIS score determined by the investigator | 4 months after initiating side 1 treatment
  Percentage of research subjects to which the investigator assigned a GAIS score to Side 1, 4 months after initiating treatment, indicating aesthetic improvement (GAIS score between 3 and 5) in relation to pre-treatment condition.
Evaluate aesthetic effect of Sculptra on skin flaccidity by comparing Side1 to Side2 by the investigator. | 4 months after initiating Side 1 treatment
  Percentage of research subjects to which the investigator determined that the treated side (Side1) is aesthetically better than the non-treated side, 4 months after initiating Side1 treatment.
Assess the aesthetic effect of Sculptra on skin flaccidity, by comparing S1 to S2 by the research subject. | 4 months after initiating side 1 treatment
  Percentage of research subjects evaluating the treated side (Side1) as aesthetically better than the non-treated side (Side2), 4 months after initiating Side1 treatment.
Assess the effect of Sculptra on dermal thickness, via high-frequency ultrasound. | 4, 6 and 12 months after initiating side 1 treatment as well as 2 and 8 months after initiating Side 2 treatment
  8.1. Variation of Side1 dermal thickness between baseline visit and 4 months after initiating treatment.
  8.2. Variation of Side1 dermal thickness between baseline visit and 6 months after initiating treatment.
  8.3. Variation of Side1 dermal thickness between baseline visit and 12 months after initiating treatment.
  8.4. Variation of Side2 dermal thickness between baseline visit and 2 months after initiating treatment.
  8.5. Variation of Side2 dermal thickness between baseline visit and 8 months after initiating treatment.
Assess the subject s discomfort with Sculptra application. | 1 year
  Mean score of subject s discomfort with Sculptra application during treatment period.
Evaluate Sculptra effect on arm circumference, 4, and 12 months after initiating Side 1 treatment | 4 and 12 months after initiating side 1 treatment
  10.1. Variation of Side1 arm circumference between baseline visit and 4 months after initiating treatment.
  10.2. Variation of Side1 arm circumference between baseline visit and 12 months after initiating treatment.
Assess investigator s satisfaction and perception of aesthetic result obtained with Sculptra. | 4, 6 and 12 months after initiating side 1 treatment as well as 6 and 8 months after initiating side 2 treatment
  11.1.Descriptive statistics of the satisfaction questionnaire and aesthetic result perception, completed by the investigator 4 months after initiating Side1 treatment.
  11.2. Descriptive statistics of the satisfaction questionnaire and aesthetic result perception, completed by the investigator 6 months after initiating Side1 treatment.
  11.3. Descriptive statistics of the satisfaction questionnaire and aesthetic result perception, completed by the investigator 12 months after initiating Side1 treatment.
  11.4. Descriptive statistics of the satisfaction questionnaire and aesthetic result perception, completed by the investigator 6 months after initiating Side2 treatment.
  11.5. Descriptive statistics of the satisfaction questionnaire and aesthetic result perception, completed by the investigator 8 months after initiating Side2 treatment.
Assess subject s satisfaction and aesthetic result perception obtained with Sculptra | 4, 6 and 12 months after initiating Side 1 treatment, as well as 6 and 8 months after initiating Side2 treatment
  12.1. Descriptive statistics of satisfaction questionnaire and aesthetic result perception, completed by the subject 4 months after initiating Side1 treatment.
  12.2. Descriptive statistics of satisfaction questionnaire and aesthetic result perception, completed by the subject 6 months after initiating Side1 treatment.
  12.3. Descriptive statistics of satisfaction questionnaire and aesthetic result perception, completed by the subject 12 months after initiating Side1 treatment.
  12.4. Descriptive statistics of satisfaction questionnaire and aesthetic result perception, completed by the subject 6 months after initiating Side2 treatment.
  12.5. Descriptive statistics of satisfaction questionnaire and aesthetic result perception, completed by the subject 8 months after initiating Side2 treatment.
Incidence, seriousness, severity and relationship of adverse events with the treatment with Sculptra | An average of 1 year
  13.1. Incidence, seriousness, severity and relationship with management of adverse events reported during study period.
  13.2. Incidence, seriousness, severity and relationship with management of adverse events of interest reported during study period.
  13.3. Incidence of treatment discontinuations due to adverse events reported during study period

CONTACTS AND LOCATIONS:
Overall Officials: Samira Yarak, Principal Investigator — Federal University of São Paulo; Marisa G Cunha, Principal Investigator — Fundacao do ABC; Doris M Hexsel, Principal Investigator — Centro Brasileiro de Estudos em Dermatologia; Alessandra Haddad, Principal Investigator — Hospital Israelita Albert Einstein
Locations (4):
- Brazil (4):
  - Centro Brasileiro de Estudos em Dermatologia, Porto Alegre, Rio Grande do Sul
  - Fundação do ABC, São Paulo, São Paulo
  - Hospital Israelita Albert Einstin, São Paulo, São Paulo
  - Universidade Federal de São Paulo - UNIFESP - UNICCO, São Paulo

IPD SHARING:
Plan to Share IPD: No